CLINICAL TRIAL: NCT06738966
Title: An International, Multi-Center, Open-label Phase I Study to Evaluate the Tolerance, Pharmacokinetics, and Anti-Tumor Effects of BL0175 Injection in Postmenopausal Female Adults With HR-positive, Locally Advanced or Metastatic Cancer
Brief Title: A Study of BL0175 Injection in Postmenopausal Female Adults With HR-positive, Locally Advanced or Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Best-Link Bioscience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL0175-102
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Ovarian Cancer; Endometrial Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BL0175 50 mg (Experimental)
  Interventions: Drug: BL0175
- BL0175 100 mg (Experimental)
  Interventions: Drug: BL0175
- BL0175 200 mg (Experimental)
  Interventions: Drug: BL0175
- BL0175 400 mg (Experimental)
  Interventions: Drug: BL0175
- BL0175 500 mg (Experimental)
  Interventions: Drug: BL0175

INTERVENTIONS:
Drug: BL0175 — BL0175 is a nano-medicine for cancer therapy. "Nano-medicine" means the tiny size of this study drug allows it to enter and concentrate into the tumor tissue. This is a new way of delivering an active drug (an estrogen receptor down regulator) for the treatment of tumor directly into tumor tissue.

SUMMARY:
The goal of this clinical trial is to learn if the investigational drug BL0175 works to treat adult postmenopausal women with hormone receptor (HR)-positive, human epidermal growth factor receptor (HER2)-negative locally advanced or metastatic breast cancer, ovarian cancer and endometrial cancer. It will also learn about the safety of BL0175. The main questions it aims to answer are:

* Does the investigational drug BL0175 is safe for participants after dosed -multiple times?
* Which is the highest safety dose of BL0175 after multiple dose?
* What medical problems do participants have when using BL0175?
* Does the investigational drug BL0175 works for participants after dosed -multiple times?

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study, be able to understand the requirements of a clinical study, and willingness to sign a written informed consent form.
2. Age ≥ 18 years.
3. HR-positive, HER2-negative (characterized by the absence of HER2 expression and the presence of ER and/or PR expression) locally advanced or metastatic breast cancer (histological or cytological proven diagnosis) in postmenopausal women with disease progression during or following endocrine therapy, or HR-positive, locally advanced or metastatic ovarian cancer or endometrial cancer in postmenopausal women that progressed during or following prior standard of care therapy.
4. Patients with at least one measurable or evaluable lesion: At least one lesion (measurable and/or non-measurable) that can be accurately assessed by CT/MRI/plain x-ray at baseline and follow up visit.

   Note: Measurable lesions cannot be selected from the following sites in principle: having received prior radiotherapy or having received other local therapy. If a target lesion at a site that has received prior radiotherapy or other local therapy is the only optional lesion, the progression of the lesion shall be confirmed by the investigator.
5. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 at screening.
6. Life expectancy period ≥ 12 weeks.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) metastases or carcinomatous meningitis.

   Note: patients with treated CNS metastases may participate in this study if the patient has completed radiotherapy or surgery for CNS metastases ≥ 4 weeks prior to study entry, and if the patient is neurologically stable ≥ 2 weeks after radiotherapy or surgery treatment (no new neurologic deficits from brain metastasis on screening clinical examination, no new findings on CNS imaging, and corticosteroids were not required within 2 weeks prior to enrollment).
2. Patients who have a history of another primary malignancy (with the exception of participants with cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of uterine cervix). A patient who has had no evidence of disease from another primary cancer for 3 or more years is allowed to participate in the study.
3. Patients whose pericardial effusion, pleural effusion or ascites remain uncontrollable after intervention.
4. Patients with a history of allogeneic transplantation of organs, bone marrow or stem cell.
5. A history of allergic or adverse response(s) to fulvestrant, or prone to allergic reactions (such as: prone to angioedema, urticaria, asthma, rash, etc.).
6. Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * New York Heart Association class III-IV for cardiac insufficiency or left ventricular ejection fraction < 50% (if the LVEF data is available).
   * Patients with poorly controlled arrhythmia: QTc interval > 480 ms calculated by Fridericia's formula, or congenital syndrome of prolonged QT interval.
   * Any of the following within 6 months prior to the enrollment: myocardial infarction, severe or unstable angina, congestive heart failure, cerebrovascular accident (including transient ischemic attack), symptomatic pulmonary embolism or other clinically significant thromboembolic disease, or coronary artery bypass graft.
   * Clinically symptomatic bradycardia as assessed by the investigator.
   * Patients with other clinically significant cardiovascular disease who were assessed as unsuitable for this study by the investigator.
7. Patients who have a known diagnosis of Human Immunodeficiency Virus (HIV) infection or HIV antibody test positive in screening.
8. Patients with active hepatitis C or chronic hepatitis B at screening ("active hepatitis" defined as HCV RNA level ≥ 200 IU/mL for hepatitis C or HBV DNA level ≥ 2000 IU/mL for hepatitis B at screening). In addition, eligible hepatitis B or hepatitis C patients must agree to antiviral treatment according to the treatment guidelines.
9. Active infections requiring antibiotic intravenous therapy within 1 weeks prior to enrollment.
10. Moderate or severe hepatic impairment (Child-Pugh class B or C).
11. Patients who have not sufficient baseline organ function and whose laboratory data meet the following criteria at enrollment [No transfusion of blood products (including platelets or red blood cells) or use of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 14 days prior to screening]:

    * Absolute Neutrophil Count (ANC) < 1.5×109/L.
    * Total bilirubin > 1.5×ULN.
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3×ULN without liver metastases or primary liver cancer. AST or ALT > 5×ULN if the patient has documented liver metastases.
    * Hemoglobin < 90 g/L.
    * Platelets < 100×109 /L.
    * Creatinine clearance < 30 mL/min.
12. Prior to first dose of the investigational product, received an antitumor drug or investigational drug at the following time intervals:

    * Chemotherapy, targeted small molecule therapy or radiotherapy (except palliative radiotherapy and the radiotherapy area do not include the proposed target lesion) ≤ 14 days. The wash-out period for TKI drugs is more than 5 half-lives could enroll for their shorter half-life.
    * Immunotherapy or cell therapy (i.e. chimeric antigen receptor T cell therapy) ≤ 28 days; Other cell therapy must be discussed with the investigators to determine eligibility.
    * Monoclonal antibodies ≤ 28 days for anticancer therapy.
    * Anti-tumor Chinese medicine which approved by the agency ≤ 14 days.
    * Immunosuppressive therapy for any reason ≤ 7 days.
    * Fulvestrant ≤ 250 days (5 half-lives).
    * All other investigational drugs or devices ≤ 28 days or 5 half-lives before the first dosing administration (whichever is shorter).
13. Bleeding constitution (e.g., diffuse intravascular coagulation [DIC], clotting factor deficiency), or long-term anticoagulant therapy (excluding antiplatelet therapy and low doses of warfarin and low molecular weight heparin).
14. Severe vascular embolism events requiring medical or surgical intervention.
15. Active autoimmune diseases that require systemic treatment (i.e. use of immunomodulators, corticosteroids, or immunosuppressive drugs).

    Note: Participants with hyperthyroidism/hypothyroidism could participate. Note: Hormone replacement therapy and symptomatic therapy (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered a form of systemic therapy and are permitted.
16. Those who have received systemic corticosteroids within 4 weeks prior to administration of BL0175 or active control (low doses of corticosteroids are excluded, such as ≤ 20 mg prednisone daily or equivalent).
17. Those who underwent major surgery within 4 weeks before enrollment, or plan to undergo major surgery during the study.
18. Has not recovered from the toxic effects of prior treatment (including prior immunotherapy) and/or complications of surgical intervention to CTCAE v5.0 ≤ 1.

    Note: Participants with stable chronic AE (≤ grade 2) that are not expected to resolve on their own (e.g., peripheral neuropathy and alopecia) are allowed.
19. Those who are determined disqualified to join clinical studies by investigator for other causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) | 0, 3, 6, 24, 48, 72, 96, 168, 240, 336 hours post first and sixth dose; before the third, fourth and fifth dose
Maximum Blood Concentration of Investigational Drug | 0, 3, 6, 24, 48, 72, 96, 168, 240, 336 hours post first and sixth dose; before the third, fourth and fifth dose
Trough Blood Concentration of Investigational Drug | 0, 3, 6, 24, 48, 72, 96, 168, 240, 336 hours post first and sixth dose; before the third, fourth and fifth dose
Half-life of Investigational Drug | 0, 3, 6, 24, 48, 72, 96, 168, 240, 336 hours post first and sixth dose; before the third, fourth and fifth dose
Progression Free Survival | From enrollment to the date of disease progress, usually of 6 months
One year survival rate | From enrollment to the time of 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No